CLINICAL TRIAL: NCT01057641
Title: A Clinical Study on the Treatment of Degenerative Lumbar Spine Stenosis With a Percutaneous Interspinous Implant in Comparison With the Best Non-operative Treatment of Lumbar Spine Stenosis
Brief Title: Study on the Treatment of Degenerative Lumbar Spine Stenosis With a Percutaneous Interspinous Implant
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: low enrollment
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Dr. Gregor Stein, Dr. med, University of Cologne
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI-DLSS
Record Dates: First submitted 2010-01-26; First posted 2010-01-27 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2016-11

CONDITIONS: Lumbar Spinal Stenosis
Keywords: PIDLSS, Spacer
MeSH Terms: conditions — Spinal Stenosis | interventions — Metered Dose Inhalers; Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Spacer (Experimental): Implantation of a percutaneously implanted interspinous device ("spacer")
  Interventions: Procedure: Spacer
- physiotherapy (Other): The control group will receive at least physiotherapy and physical therapy (e.g. massage and fango). Under inpatient conditions therapy will last for seven days. After discharge physical therapy has to be continued for 5 weeks. A schedule will ensure the consistency of the physical therapy. The inpatient-treatment can be repeated every 6 months if necessary.
  Interventions: Other: physiotherapy

INTERVENTIONS:
Procedure: Spacer — Implantation of a percutaneously implanted interspinous device (spacer)
  Other Names: PIDLSS
  Arms: Spacer
Other: physiotherapy — physiotherapy
  Other Names: PIDLSS
  Arms: physiotherapy

SUMMARY:
Neurogenic intermittent claudication is a specific symptom complex occurring in patients with lumbar spinal stenosis. Characteristic of this disease is the occurrence of increasing leg, buttock or groin pain with or without lower back pain when walking a certain distance or reclining. Bending forward or sitting leads to a rapid pain relief. Lumbar spinal stenosis is defined as a reduction of the diameter of the spinal canal. The mechanism leading to stenosis is a remodeling and overgrowth of the spinal canal with osteophyte formation. Any loss of tissue or decrease of the disc height results in a relative laxity of the ligament structures and accelerates the degeneration of the spinal joints. As a therapy option, conservative therapy with oral analgesics and physical therapy is considered. This treatment can be intensified by adding epidural pain treatment. Is the conservative treatment not successful surgical intervention is necessary. In patients over 65 years of age operative decompression of the lumbar spinal stenosis constitutes the most common surgical operation of the spine. A relatively new therapy alternative is the interspinous process decompression (IPD). Studies have shown that the IPDs prevent narrowing of the spinal canal and neural foramens. The study is intended as a randomised, monocentre study to investigate the safety and the benefit of a minimally invasive percutaneous IPD-device in comparison with the best non-surgical operative treatment of lumbar spinal stenosis.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female over 50 years of age
2. One, two, or three segment degenerative lumbar spinal stenosis (DLSS)
3. Symptoms of radiographically confirmed DLSS like leg, buttock, or groin pain with or without back pain and absence of a peripheral motoric deficit
4. Pain relief in inclination or sitting
5. Ability to walk over a distance of 50 m
6. Unsuccessful conservative therapy for 3 months under outpatient conditions
7. Informed consent

Exclusion Criteria:

1. Fixed motoric deficit
2. Cauda equina syndrome
3. Previous surgery of the lumbar spine
4. Severe osteoporosis of the vertebrae and/or of the hip
5. Spondylolisthesis more severe than Meyerding I (on scale of I-IV)
6. Metastasis of the vertebrae
7. Mentally disabled persons

Ages: 50 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-03; Primary Completion 2016-05 (Actual); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Changes in subscores for bodily pain and physical function on SF-36 | baseline, 6 months

SECONDARY OUTCOMES:
Symptoms severity by applying the Zurich Claudication Questionaire (ZCQ) | baseline, 6 months
Physical function by applying ZCQ | baseline, 6 months
Post-treatment patient satisfaction by applying ZCQ | baseline, 6 months
General health status (Quality of life) by applying SF-36 | baseline, 6 months
Measurement of walking distance | baseline, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Kaulhausen, MD, Principal Investigator — University Hospital of Cologne
Locations (2):
- Germany (2):
  - University Hospital Cologne, Cologne, North Rhine-Westphalia
  - University Hospital of Cologne, Cologne